CLINICAL TRIAL: NCT01849939
Title: Reduced Intensity Conditioning Allogeneic Transplantation for CLL With Preemptive MDR Management (ICLL 03 RICAC-PMM)
Brief Title: Eradication of Residual Disease by Preemptive Immunointervention After Allogeneic Hematopoietic Stem Cells Transplantation in Chronic Lymphocytic Leukemia
Acronym: RICAC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Pierre Fabre Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHU-0150; 2011-A00906-35
Record Dates: First submitted 2013-03-12; First posted 2013-05-09 (Estimated); Last update posted 2013-05-09 (Estimated); Status verified 2013-05

CONDITIONS: Chronic Lymphocytic Leukemia; Lymphocytic Lymphoma
Keywords: Allogeneic transplantation of hematopoietic stem cells transplantation; Chronic Lymphocytic Leukemia; Donor Lymphocyte Injection; Preemptive immunointervention
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

ARMS (1):
- Fludarabin (Experimental)
  Interventions: Drug: Fludarabin (post-allograft immunosuppressive therapy modulation and DLI Mononuclear cells from allogenic blood)

INTERVENTIONS:
Drug: Fludarabin (post-allograft immunosuppressive therapy modulation and DLI Mononuclear cells from allogenic blood)

SUMMARY:
Usually Chronic lymphocytic leukemia (CLL) is a disease of the elderly patients. However, the diagnosis in young patients become more frequently with poor prognosis. The identification of new prognostic factors permits early determination of the high risk population and provide them the therapeutic intensification. Allogeneic transplantation of hematopoietic stem cells transplantation (AHSCT) allows to long-term remission and in some cases complete and definitive eradication of the disease. After chemotherapy or antibodies, the Minimal Residual Disease (MRD) negativity is associated with better disease-free survival. MRD negativity occurs in some patients with the appearance of GVHD, stopping the immunosuppression or after donor lymphocyte injection (DLI). The negativity of MRD in the first year post-transplant is correlated with better progression-free survival or overall survival (Dreger 2010, Farina 2009, Caballero 2005, Algrin, 2011). So, MRD negativity may be an objective after AHSCT. The aim of this prospective study is to evaluate a standardized preemptive immunointervention of post-allograft immunosuppressive therapy modulation and DLI administration according to MRD level. The objective is to obtain MRD negativity at 12 months after AHSCT.

DETAILED DESCRIPTION:
Patients will receive AHSCT with Fludarabine-Busulfan based conditioning :

* Fludarabine : 30 mg/m2/day - from Day-6 to Day-2
* Busulfan IV : 3.2 mg/kg/day - on Day-5 and Day-4
* ATG (Anti-thymocyte Globulin) : 2.5 mg/kg/day on Day-2 and Day-1

Preemptive immunointervention post AHSCT consists in reduce immunosuppressive treatment more or less associated with DLI according to :

* the presence or absence of severe Graft versus host disease (GVHD) (acute grade 2 and / or chronic)
* the presence or absence of a response on criteria of response IWCLL
* Getting or not a blood MRD negative (<-10 ^ -4) evaluated by flow cytometry

ELIGIBILITY:
Inclusion Criteria:

* Patients with CLL (Matutes score 4 or 5) stages A, B, C with evolution criteria according IWCLL 2008 or lymphocytic lymphoma with severity criteria (EBMT criteria) which indicated allograft (deletion 17p) and requiring treatment
* Age: 18-70 years
* At least one of the following criteria of poor prognosis (EBMT recommendations - Dreger 2007)

  1. No response or relapse within 12 months of treatment with purine analogues (including "fludarabine refractory" i.e patients in response <PR and / or relapse within 6 months after at least 2 courses of Fludurabine)
  2. relapse within 24 months after combination therapy including purine analogs or autograft, with indication of new start of treatment
  3. Mutation/deletion 17p13 (p53) with indication for treatment
* Partial response (PR) or complete response (CR) at the last treatment (IWCLL 2008)
* Residual mass <5 cm (clinical and CT scan)
* Identical intrafamilial donor HLA (or with a mismatch) or in the absence of family donor, an unrelated donor 10/10 for HLA A, B, C, DR, DQ and is committed to giving DLI (see consent form donor)
* Sorror score comorbidity: ≤ 2
* Written informed consent
* Member or beneficiary of a social security system

Exclusion Criteria:

* Richter Syndrome
* Usual contraindications for realisation of allogeneic transplantation including
* Uncontrolled bacterial, viral or fungal infection
* Pregnancy or lactating women
* Cardiac contraindication : Cardiac ejection fraction <50%
* Pulmonary contraindication : DLCO <50%
* Renal contraindication : Creatininine clearance <30 ml / min
* Hepatic contraindication : AST and / or ALT and / or total bilirubine> 2 N except Gilbert disease or localisation specific LLC
* HIV positivity
* Cancer evolution or de novo occurred in the previous 5 years except basal cell cancer skin or carcinoma in situ of the cervix of uterus
* Affection psychiatric disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2012-09; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
MRD(Minimal Residual Disease) negativity level | 12 months after AHSCT(Allogenic Transplantation of Hematopoietic Stem Cells Transplantation)

SECONDARY OUTCOMES:
Incidence of relapses progression | at 12 months
Incidence of toxic deaths | at 12 months
Incidence of GVHD (acute and chronic) | at 12 months
Survival (progression free survival, overall survival, survival without treatment) | at 12 months
Post-transplant chimerism (total blood and lymphoid T lymphocyte populations) | baseline; 1, 2, 3, 6 and 12 months
Incidence of infectious complications and severity | at 12 months
  The aim of this prospective study is to evaluate a standardized preemptive immunointervention of post-allograft immunosuppressive therapy modulation and DLI administration according to MRD level. The objective is to obtain MRD negativity at 12 months after AHSCT

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Tournilhac, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France